CLINICAL TRIAL: NCT01165879
Title: Measuring Uterine Electrical Activity Throughout Pregnancy and Labor Measuring Uterine Electrical Activity Throughout Pregnancy and Labor
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: OB-Tools Ltd. (Industry)
Responsible Party: Dr. Tal Biron Shental, Meir Medical Center
Other Study IDs: HTA5347
Record Dates: First submitted 2010-07-18; First posted 2010-07-20 (Estimated); Last update posted 2011-06-10 (Estimated); Status verified 2010-07

CONDITIONS: Pregnancy
Keywords: Pregnancy; Term; Preterm; Uterine Contractions
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The EUM100pro (Electrical Uterine Monitor)is a uterine contraction monitor which measures uterine contractions based on the electrical activity of the uterine muscle.The study will compare the EUM100pro measurements to the already existing uterine contractions monitors (tocodynamometer and Intra Uterine Pressure Catheter) in pregnant women with complaints of uterine contractions.

DETAILED DESCRIPTION:
The main objective of the study is to demonstrate that the EUM100pro is as good as the current methods for monitoring pregnancy in labor (tocodynamometer, IUPC) in measuring uterine contractions. This will be performed by measuring the expectancy of time differences between the tocodynamometer/IUPC and the EUM in the beginning, end, peak and duration of each contraction. A good correlation will be 0.9 and significance of 95%.

100 women will be recruited to the study. The measurement with the EUM100pro will not interfere with the usual clinical care, meaning- the EUM100pro will be used in addition to the standard care and monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Women at term with complaint of uterine contractions at Meir Medical Center
* Women at preterm with complaint of uterine contractions at Meir Medical Center.
* Women at gestational age >24 weeks
* Subjects who understood, agreed and signed the informed consent form

Exclusion Criteria:

* Subjects who refused to sign the informed consent form
* Abnormal fetal heart rate recording at admittance
* Subjects with indications for immediate delivery
* Subjects younger than 18 years of age
* Subjects at gestational age <24 weeks

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Pergnant women which are admitted to Meir Medical Center with complaints of uterine contractions starting.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2010-05; Primary Completion 2012-05 (Estimated)

PRIMARY OUTCOMES:
The study primary outcome is to demonstrate that the EUM100pro uterine contractions measurements is as good as the current methods for monitoring pregnancy in labor (tocodynamometer, IUPC). | two years
  The primary outcome will be measured by correlation of timing of :peak display in beginning, during and end of peak in the EUM100pro versus the timing of the peak display in beginning, during and the end tocodynamometer and or IUPC peak.
To evaluate patient safety | one year
  Measurements of device related adverse events throughout the study.

SECONDARY OUTCOMES:
Correlation of uterine contractions intensity between EUM100pro and Intra Uterine Pressure Catheter measurements. | one year
  The secondary outcome will investigate a correlation between the intensity/peak of contraction of mechanical contraction as measured by Intra Uterine pressure catheter and the intensity/peak of contraction of electrical activity as measured by the EUM exists.
To evaluate usability of the EUM100pro | one year
to evaluate whether a fetal ECG can be exctraced from the electrical signal of the uterus. | one year
  The electrical signal recorded from the abdomen thechnically contain the uterine muscle electrical activity but also the electrical signal from the fetal ecg.

CONTACTS AND LOCATIONS:
Overall Officials: Tal Shental Biron, MD, Principal Investigator — Meir Hospital
Locations (1):
- Meir Medical Center, Kfar Saba, Israel